CLINICAL TRIAL: NCT03864354
Title: The Immediate, Intermediate, and Long-Term Effects of Osteopathic Manipulative Treatment on Pulmonary Function in Adults With Asthma
Brief Title: Asthma and Osteopathic Manipulative Treatment
Status: Completed | Type: Observational
Sponsor: Des Moines University (Other)
Responsible Party: Sponsor
Other Study IDs: Asthma and OMT
Record Dates: First submitted 2019-02-20; First posted 2019-03-06 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Asthma
Keywords: osteopathic manipulative medicine; Spirometry; Respiratory; OMM; OMT; osteopathic manual medicine; osteopathic manipulative treatment; osteopathic manual treatment
MeSH Terms: conditions — Asthma | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Participants were adults with a diagnosis of asthma, treated using a standardized Osteopathic Manipulative Treatment protocol.
  Interventions: Procedure: Osteopathic Manipulative Treatment

INTERVENTIONS:
Procedure: Osteopathic Manipulative Treatment — Osteopathic Manipulative Treatment (OMT) is a cost-effective, noninvasive treatment that is used to optimize the body's structure and function. By improving the biomechanical, autonomic, and circulatory mechanisms involved in the disease process of asthma, OMT can help maximize respiratory function. The specific OMT protocol used in this study included the following: supine OA joint myofascial release (MFR), supine cervical spine Still technique, supine thoracic inlet MFR, supine rib raising soft tissue, supine rib MFR, supine abdominal diaphragm MFR, seated thoracic spine Still technique, and seated posterior rib Still technique. Treatments were performed by Predoctoral Osteopathic Manipulative Medicine (OMM) Fellows at Des Moines University (DMU) and supervised and checked by one of two board-certified OMM/NMM physicians from the OMM Department at DMU. The treatment lasted an average of 21 minutes and repeated three times, spaced one week apart.

SUMMARY:
The effect of Osteopathic Manipulative Treatment (OMT) has been studied in adult patients with chronic obstructive pulmonary disease (COPD) and children with asthma, however, to the authors' knowledge, no current studies have evaluated the non-immediate effects of OMT on pulmonary function in adults with chronic asthma using spirometry. The objective of the current study was to quantify the immediate, intermediate, and long-term effects of OMT on adult patients with a history of asthma. The quantitative effects were measured with a spirometry device and include the forced expiratory volume in one second (FEV1), the forced vital capacity (FVC), the FEV1/FVC ratio, and the peak expiratory flow (PEF). These four values are used clinically in the diagnosis and management of asthma. The long-term, subjective effects were measured via the Asthma Quality of Life Questionnaire with Standardized Activities (AQLQ(S)).

The study was conducted over a period of eight weeks. During week 0, participants completed the initial AQLQ and performed baseline spirometry testing. During weeks 1, 2, and 3 of the study, a standard OMT protocol was performed on each participant, followed by spirometry testing to measure the immediate effect. Spirometry testing was then performed again three days after each treatment to measure the intermediate effect of OMT. During week 7, participants completed the post-OMT AQLQ(S) and performed spirometry testing once more to measure the long-term effects of OMT. The OMT protocol performed on each patient included treatments to address somatic dysfunctions of the head, cervical spine, thoracic spine, ribs, and respiratory diaphragm. The authors hypothesized that OMT would improve pulmonary function, both subjectively and objectively. The authors predicted an increased overall mean AQLQ(S) score as well as an increased mean score within each domain, including symptoms, activity limitations, emotional function, and environmental stimuli. The authors also predicted a significant increase in the mean FEV1/FVC ratio, and PEF three days after each OMT session and a significant increase four weeks after the final OMT session, but no increase immediately after OMT.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* previously diagnosed with asthma

Exclusion Criteria:

* Current smoker
* Diagnosed with any other respiratory disease besides asthma
* Receiving OMM from a licensed physician, chiropractic treatment, or massage therapy for 30 days prior to and during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants included members of the Des Moines University community.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume in one second (FEV1) measured in liters by a spirometer | Measured during weeks 0 (at baseline), 1, 2, 3, and 7 of the study to assess the change over time. During weeks 1, 2, and 3, spirometry was performed immediately after the OMT protocol was completed as well as three days later.
Asthma Quality of Life Questionnaire with Standardized Activities (AQLQ(S)) | Participants completed the survey at baseline and four weeks after the last treatment to compare the change.
  The AQLQ asks about a participant's past 2 weeks as they relate to their symptoms, activity limitations, emotional function, and environmental stimuli. Each item is a 7-point Likert scale, with 1 being severely impaired and 7 not impaired at all.
Forced vital capacity (FVC) measured in liters by a spirometer | Measured during weeks 0 (at baseline), 1, 2, 3, and 7 of the study to assess the change over time. During weeks 1, 2, and 3, spirometry was performed immediately after the OMT protocol was completed as well as three days later.
Forced expiratory flow in one second to forced vital capacity ratio (FEV1/FVC ratio) by a spirometer | Measured during weeks 0 (at baseline), 1, 2, 3, and 7 of the study to assess the change over time. During weeks 1, 2, and 3, spirometry was performed immediately after the OMT protocol was completed as well as three days later.
Peak expiratory flow (PEF) measured in liters per minute by a spirometer | Measured during weeks 0 (at baseline), 1, 2, 3, and 7 of the study to assess the change over time. During weeks 1, 2, and 3, spirometry was performed immediately after the OMT protocol was completed as well as three days later.

CONTACTS AND LOCATIONS:
Locations (1):
- Des Moines University, Des Moines, Iowa, United States

IPD SHARING:
Plan to Share IPD: Undecided
The investigator's study is a pilot study. If members of the OMM department at DMU choose to continue researching the effects of OMT on asthma in the future, then the data collected in the present study would be shared with those department members.

REFERENCES:
- [Background] Bockenhauer SE, Julliard KN, Lo KS, Huang E, Sheth AM. Quantifiable effects of osteopathic manipulative techniques on patients with chronic asthma. J Am Osteopath Assoc. 2002 Jul;102(7):371-5; discussion 375. PMID 12138951
- [Background] McCracken JL, Veeranki SP, Ameredes BT, Calhoun WJ. Diagnosis and Management of Asthma in Adults: A Review. JAMA. 2017 Jul 18;318(3):279-290. doi: 10.1001/jama.2017.8372. PMID 28719697
- [Background] Thiadens HA, De Bock GH, Van Houwelingen JC, Dekker FW, De Waal MW, Springer MP, Postma DS. Can peak expiratory flow measurements reliably identify the presence of airway obstruction and bronchodilator response as assessed by FEV(1) in primary care patients presenting with a persistent cough? Thorax. 1999 Dec;54(12):1055-60. doi: 10.1136/thx.54.12.1055. PMID 10567623
- [Background] Guiney PA, Chou R, Vianna A, Lovenheim J. Effects of osteopathic manipulative treatment on pediatric patients with asthma: a randomized controlled trial. J Am Osteopath Assoc. 2005 Jan;105(1):7-12. PMID 15710659
- [Background] Noll DR, Degenhardt BF, Johnson JC, Burt SA. Immediate effects of osteopathic manipulative treatment in elderly patients with chronic obstructive pulmonary disease. J Am Osteopath Assoc. 2008 May;108(5):251-9. PMID 18519835
- [Background] Henderson AT, Fisher JF, Blair J, Shea C, Li TS, Bridges KG. Effects of rib raising on the autonomic nervous system: a pilot study using noninvasive biomarkers. J Am Osteopath Assoc. 2010 Jun;110(6):324-30. PMID 20606239
- [Background] Juniper EF, Guyatt GH, Willan A, Griffith LE. Determining a minimal important change in a disease-specific Quality of Life Questionnaire. J Clin Epidemiol. 1994 Jan;47(1):81-7. doi: 10.1016/0895-4356(94)90036-1. PMID 8283197
- See also: Asthma Care Quick Reference: Diagnosing and Managing Asthma — https://www.nhlbi.nih.gov/files/docs/guidelines/asthma_qrg.pdf
- See also: CDC's Most Recent Asthma Data — https://www.cdc.gov/asthma/most_recent_data.htm

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-08): https://cdn.clinicaltrials.gov/large-docs/54/NCT03864354/Prot_SAP_000.pdf